CLINICAL TRIAL: NCT03970525
Title: A Comparison of Venturi and Peristaltic Based Phacoemulsification in Femtosecond Laser Cataract Surgery
Brief Title: Venturi and Peristaltic Based Phacoemulsification in Femtosecond Laser Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Wendell Scott (Other)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Wendell Scott, MD, Ophthalmologist, Mercy Research
Organization: Mercy Research (Other)
Other Study IDs: 19-082
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Venturi pump: This cohort will receive femtosecond laser cataract surgery with Venturi pump.
  Interventions: Device: Venturi pump
- Peristaltic vacuum pump: This cohort will receive femtosecond laser cataract surgery with peristaltic pump.
  Interventions: Device: Peristaltic vacuum pump

INTERVENTIONS:
Device: Venturi pump — The venturi pump makes use of the venturi effect to create a vacuum. The venturi effect creates a vacuum by the flow of a fluid, typically air, over an opening. In many phacoemulsification machines, this requires nitrogen tanks or a self-contained air compressor. The vacuum level is created within a rigid drainage cassette, to which the phaco aspiration tubing is connected. Since there is no milking of the aspiration line, the phaco tubing can be made rigid with low compliance.
  Groups: Venturi pump
Device: Peristaltic vacuum pump — The peristaltic pump uses rollers to compress the phacoemulsification outflow tubing in a peristaltic manner, thereby creating flow and vacuum. The compression of the rollers on the tubing with the rotation of the pump physically moves fluid and creates a continuous "milking" action on the fluid column, The phaco machine can directly control this flow level, hence the term flow based, however, the preset vacuum level is only achieved once there is occlusion of the outflow line, typically at the phaco needle tip with cataract material.
  Groups: Peristaltic vacuum pump

SUMMARY:
This study will compare two methods of vacuum (peristaltic or venturi) commonly used during the removal of a femtosecond treated cataract. The investigators will observe which method uses less energy, is gentler on the eye, reduces corneal swelling and if the vision recovers faster with one method compared to the other.

DETAILED DESCRIPTION:
This is an open, prospective, randomized study to evaluate efficiency and outcomes of femtosecond laser cataract surgery with phacoemulsification performed with one of two standard vacuum systems.

It is estimated that the duration of study participation will be up to 24 months.

There will be randomization to 1 of 2 groups. Both eyes of each subject will be enrolled in the study. The first eye will be randomized to either the Venturi or peristaltic-based vacuum pump. The second eye will then receive the other type of vacuum pump for that procedure.

Study Phases:

Pre-operative Visit Procedure Post-operative Follow up The subject will be seen 1 day, 5-10 days, and 90 days following the procedure.

Surgical Procedure

* The cataract removal procedure will be performed under sterile technique and according to standard procedures. The femtosecond laser treatment will be followed by phacoemulsification removal of the cataract and implantation of an intraocular lens.
* Peri-operatively, subjects will be treated with a regimen of antibiotic, steroid and nonsteroidal anti-inflammatory eye drops per standard of care.
* All surgeries will be performed by the same experienced surgeon/principal investigator using the Catalys® SYSTEM femtosecond laser platform and WHITESTAR SIGNATURE® PRO Phacoemulsification System.
* Phacoemulsification Settings:

  * For Venturi pump: 600 mmHg vacuum
  * For Peristaltic-based pump: 600 mmHg vacuum and aspiration flow of 50 mL/min
  * Other settings: ultrasound energy application parameters will be the same for the two groups

Study Procedures

* The study will include routine cataract pre-operative testing with Nidek OPD, Galilei G4, and IOLMaster, and repeated at the post-op visits. An endothelial cell count of the cornea will be performed at the pre-operative visit and at the 90 day follow up visit.
* Subjects will be randomized to phacoemulsification settings of Venturi vacuum of 600 mmHg or peristaltic vacuum of 600 mmHg and aspiration flow of 50 mL/min. All other phacoemulsification settings will be identical. The laser settings will be based on the grade of cataract only and will not be altered for this study.
* The phacoemulsification time, energy Ellips FX EFX, and average phacoemulsification energy will be recorded. The laser procedure time and total procedure time will be recorded. Complications will be recorded. Additional patient characteristics will also be recorded.
* Pre-Operative Visit:

  * Nidek Refractive Power/Corneal Analyzer OPD-Scan, Galilei G4 Corneal Topography, IOLMaster 700 keratometry (standard of care)
  * Complete eye examination (standard of care)
  * Brightness Acuity Test (BAT) (standard of care)
  * Review and confirm eligibility (research)
  * Informed Consent for study (research)
  * Randomization (research)
  * Endothelial Cell Count (research)
  * Medical Record Review (research)
* Surgical Procedure (Day 0) (standard of care)

  * Medical Record Review (research)
  * Adverse Event Assessment (research)
* Post-operative Visit 1 (Day 1):

  * Eye exam to include uncorrected and pinhole visual acuity, Intraocular pressure (IOP) and slit-lamp exam (standard of care)
  * Galilei G4 Corneal Topography, IOLMaster 700 keratometry (standard of care)
  * Medical Record Review (research)
  * Adverse Event Assessment (research)
* Post-operative Visit 2 (Day 5-10):

  * Eye exam to include uncorrected and best corrected visual acuity, Pinhole visual acuity, IOP, and slit-lamp exam (standard of care)
  * Nidek Refractive Power/Corneal Analyzer OPD-Scan, Galilei G4 Corneal Topography, IOLMaster 700 keratometry (standard of care)
  * Medical Record Review (research)
  * Adverse Event Assessment (research)
* Post-operative Visit 3 (Day 60-90 days):

  * Eye exam to include uncorrected and best corrected visual acuity, Pinhole visual acuity, IOP, and slit-lamp exam (research)
  * Nidek Refractive Power/Corneal Analyzer OPD-Scan, Galilei G4 Corneal Topography, IOLMaster 700 keratometry (research)
  * Endothelial Cell Count (research)
  * Medical Record Review (research)
  * Adverse Event Assessment (research)
* Unscheduled Visit:

  * A medical record review and an adverse event assessment will be performed at any unscheduled visit.
  * Additional evaluations will be completed at the discretion of the Principal Investigator based on the subject's presenting complaint.

Statistical Analysis

Sample Size and Power:

· The study aims to enroll 250 study subjects for a total of 500 eyes with bilateral grade 1-3 nuclear sclerotic cataracts who will be undergoing planned femtosecond laser cataract surgery.

Statistical Methods:

· The statistical analysis plan will include use of descriptive statistics and statistical tests including unpaired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 22-90 yrs
* Diagnosis of senile cataract
* Grade 1-3 Nuclear sclerosis
* Cataract removal required for both eyes
* Scheduled for femtosecond laser cataract surgery at Mercy Surgery Center or Mercy National Eye Center in Springfield, MO

Exclusion Criteria:

* Diagnosis of Fuch's dystrophy
* Presence of cornea scars
* Planned laser astigmatism treatment
* Diagnosis of pseudoexfoliation
* History of direct ocular trauma with secondary iris or lens trauma
* Presence of grade 4 cataracts
* History of previous eye surgery
* Severe glaucoma or retina disease impairing vision
* Planned surgery that is will be combined with other surgical eye procedures

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * The study aims to enroll 250 study subjects for a total of 500 eyes with bilateral grade 1-3 nuclear sclerotic cataracts who will be undergoing planned femtosecond laser cataract surgery.
  * The study will include adults undergoing femtosecond laser cataract surgery with grade 1-3 nuclear sclerotic cataracts.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Phacoemulsification energy required during femtosecond laser cataract surgery procedure | Intraoperative Visit
  Phaco EFX (the effective phaco time with a specific coefficient for the transversal movement of the phaco tip- expressed in seconds.)
Duration of ultrasound time required during femtosecond laser cataract surgery procedure | Intraoperative Visit
  Total ultrasound time - measured in seconds
Phacoemulsification power required during femtosecond laser cataract surgery procedure | Intraoperative Visit
  Average power - measured in percentage
Duration of microscope time required during femtosecond laser cataract surgery procedure | Intraoperative Visit
  Microscope time - measured in seconds intraoperatively
Duration of laser time required during femtosecond laser cataract surgery procedure | Intraoperative Visit
  Laser time - measured in seconds intraoperatively

SECONDARY OUTCOMES:
Uncorrected visual acuity among subjects who underwent femtosecond laser cataract surgery procedure | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  1) Uncorrected Visual Acuity using the Snellen Eye Chart
Best Corrected Visual Acuity among subjects who underwent femtosecond laser cataract surgery procedure | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  Best Corrected Visual Acuity using the Snellen Eye Chart
Pinhole Visual Acuity among subjects who underwent femtosecond laser cataract surgery procedure | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  Pinhole visual acuity using pinhole technique and the Snellen eye chart
Presence of corneal edema as assessed by intra-ocular pressure | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  Measured in mmHg using an applanation tonometer
Presence of corneal edema as assessed by slit lamp examination | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  The examiner will use a slit lamp microscope to evaluate the eye structures and intra-ocular pressure
Measure of the corneal endothelium | This test will be done Pre-operatively and Post op 60-90 day visit
  Endothelial Cell Count will be evaluated by Konan Specular Microscopy
Central corneal thickness as measured by IOLMaster Biometry | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  IOL Master Biometry directly measures the corneal thickness by OCT
Central corneal thickness as measured by Galilei G4 Biometry | This test will be done Pre-operatively and at Post op day 1, Post op day 5-10, and Post op day 60-90
  Galilei G4 measures central corneal thickness

OTHER OUTCOMES:
Adverse Events | 90 days
  Adverse Events will be recorded an monitored for each group and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Wendell J Scott, MD, Principal Investigator — Mercy Hospital
Locations (1):
- Mercy Clinic Eye specialists, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Zhao J, Xu J, Zhang J. Evaluation of the effectiveness of combined femtosecond laser-assisted cataract surgery and femtosecond laser astigmatic keratotomy in improving post-operative visual outcomes. BMC Ophthalmol. 2018 Jul 3;18(1):161. doi: 10.1186/s12886-018-0823-1. PMID 29970039
- [Background] Day AC, Smith PR, Tang HL, Aiello F, Hussain B, Maurino V, Marshall J, Saleh GM. Surgical efficiency in femtosecond laser cataract surgery compared with phacoemulsification cataract surgery: a case-control study. BMJ Open. 2018 Feb 17;8(2):e018478. doi: 10.1136/bmjopen-2017-018478. PMID 29455164
- [Background] Basic Principles of Phacoemulsification and Fluid Dynamics. Retrieved from https://www.aao.org/focalpointssnippetdetail.aspx?id=fde87039-2700-4d45-808a-9af6226a983d
- [Background] 5. Peristaltic and Venturi Fluid Pumps. Retrieved from https://www.aao.org/focalpointssnippetdetail.aspx?id=42e35231-7641-4190-b0cd-7ffdc1b8de74
- [Background] DeMill DL, Zaugg BE, Pettey JH, Jensen JD, Jardine GJ, Wong G, Olson RJ. Objective comparison of 4 nonlongitudinal ultrasound modalities regarding efficiency and chatter. J Cataract Refract Surg. 2012 Jun;38(6):1065-71. doi: 10.1016/j.jcrs.2011.12.040. PMID 22624907
- [Background] Conrad-Hengerer I, Hengerer FH, Schultz T, Dick HB. Effect of femtosecond laser fragmentation on effective phacoemulsification time in cataract surgery. J Refract Surg. 2012 Dec;28(12):879-83. doi: 10.3928/1081597X-20121116-02. PMID 23231739
- [Result] 1. Jacobs, DS. (2019). Cataract in Adults. In T.W. Post, J. Trobe & J. Givens (Eds.), UpToDate. Available from https://www.uptodate.com/contents/cataract-in-adults?search=cataract&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1
- [Derived] Scott RA, Holtmeyer CJ, Parker TM, Willis JK, Scott WJ, Olson RJ. Efficiency of venturi vs peristaltic-based phacoemulsification in femtosecond laser cataract surgery. J Cataract Refract Surg. 2025 May 1;51(5):382-387. doi: 10.1097/j.jcrs.0000000000001618. PMID 39853262